CLINICAL TRIAL: NCT02763384
Title: A Phase IIa Study of BL-8040 in Combination With Nelarabine for Relapsed or Refractory T-Acute Lymphoblastic Leukemia/ Lymphoblastic Lymphoma
Brief Title: BL-8040 and Nelarabine for Relapsed or Refractory T-Acute Lymphoblastic Leukemia/ Lymphoblastic Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Leukemia and Lymphoma Society (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201606146; 2P50CA171963-06 (NIH)
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Results first posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: T-Acute Lymphoblastic Leukemia; Adult T Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — 4-fluorobenzoyl-TN-14003; nelarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1: BL-8040 and Nelarabine (Experimental): * Cycle 1: BL-8040 subcutaneous daily from Day 1 to Day 6 and nelarabine intravenously over 2 hours on Days 2, 4, and 6
  * Cycles 2-4: BL-8040 subcutaneous daily from Day 1 to Day 5 and nelarabine intravenously over 2 hours on Days 1, 3, and 5
  * Treatment may be repeated every 21 days for up to 4 cycles
  Interventions: Drug: BL-8040; Drug: Nelarabine

INTERVENTIONS:
Drug: BL-8040
Drug: Nelarabine
  Other Names: Arranon

SUMMARY:
The outcome of patients with relapsed or refractory adult T-acute lymphoblastic leukemia (T-ALL) and the related disease T-lymphoblastic lymphoma (T-LBL) is extremely poor with 30% of the patients responding to first salvage therapy and long-term survival of only 10%. Therefore, novel therapies for patients with relapsed/refractory T-ALL/LBL represent an unmet clinical need.

Recent data provide strong evidence that CXCR4 signaling plays a major role in T-cell leukemia cell maintenance and leukemia initiating activity, and targeting CXCR4 signaling in T-ALL cells reduces tumor growth in an animal model. In this study, the investigators propose that the addition of BL-8040 to nelarabine as a salvage therapy for patients with relapsed/refractory T-ALL/LBL will result in a higher complete remission (CR) rate than nelarabine alone without an increase in toxicity and will allow patients to proceed to a potentially curative allogeneic hematopoietic cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T-acute lymphoblastic leukemia/ lymphoblastic lymphoma according to WHO criteria which has relapsed or is refractory to chemotherapy.
* Peripheral blood lymphoblasts ≤ 50,000 mcL. Hydroxyurea and/or leukapheresis is permitted to reduce the peripheral blast count prior to enrollment and treatment.
* Age ≥ 18 years
* ECOG performance status ≤ 2.
* Adequate organ function defined as:

  * Calculated creatinine clearance ≥ 50 ml/min using the Cockroft-Gault formula
  * AST, ALT, total bilirubin ≤ 2 x institutional ULN except for Gilbert's disease or when in the opinion of treating physician elevated levels are due to direct involvement of leukemia (e.g., hepatic infiltration or biliary obstruction due to leukemia), in which case ALT and AST may be elevated up to ≤ 5 x IULN.
* Women of childbearing potential and men must agree to use adequate contraception with a highly effective method (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Abstinence is acceptable if this is the established and preferred contraception for the subject.
* Female subjects must have a negative urine or serum pregnancy test within 72 hours prior to start of study treatment if of childbearing potential or be of non-childbearing potential. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the subject to be eligible. Non-childbearing potential is defined as:

  *≥ 45 years of age and has not had menses for > 2 years
  * Amenorrheic for > 2 years without a hysterectomy and oophorectomy and a FSH value in the postmenopausal range upon pretrial (screening) evaluation
  * Post-hysterectomy, oophorectomy, or tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Previous treatment with nelarabine for relapsed or refractory disease.
* Pregnant or nursing.
* Received any other investigational agent or systemic cytotoxic chemotherapy within the preceding 2 weeks.
* Active CNS involvement with leukemia
* Active HIV or hepatitis B or C infection.
* Any medical condition which, in the opinion of the clinical investigator, would interfere with the evaluation of the patient. Subjects with a clinically significant or unstable medical or surgical condition or any other condition that cannot be well-controlled by the allowed medications permitted in the study protocol that would preclude safe and complete study participation, as determined by medical history, physical examinations, laboratory tests, and according to the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey L Uy, M.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: BL-8040 and Nelarabine
Started | 12
Completed | 10
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Rapid decline - went on hospice | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1: BL-8040 and Nelarabine
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 30 [20 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Regimen as Measured by Number of Participants With Adverse Events
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all adverse event reporting.
Time Frame: Up to 30 days after completion of treatment (median follow-up of 51.5 days, full range 24-120 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: BL-8040 and Nelarabine
Number analyzed (Participants) | 12
Participants
  Grade 3-5 white blood cell increased post BL-8040 injection | 1
  Grade 1-2 lymphadenopathy worsening | 1
  Grade 3-5 leukocytosis | 1
  Grade 1-2 infarct | 1
  Grade 1-2 chest pain - cardiac | 2
  Grade 1-2 pericardial effusion | 1
  Grade 1-2 sinus bradycardia | 2
  Grade 1-2 sinus tachycardia | 3
  Grade 1-2 tinnitus | 1
  Grade 3-5 abdominal pain at study drug injection site | 1
  Grade 1-2 constipation | 2
  Grade 1-2 diarrhea | 2
  Grade 3-5 diarrhea | 1
  Grade 1-2 gastrointestinal hemorrhage | 1
  Grade 1-2 mucositis oral | 1
  Grade 1-2 nausea | 1
  Grade 1-2 oral hemorrhage | 1
  Grade 1-2 vomiting | 4
  Grade 1-2 "feeling funny" post transfusion | 1
  Grade 1-2 biopsy pain | 1
  Grade 1-2 catheter pain from replacement | 1
  Grade 3-5 disease progression | 1
  Grade 1-2 pain at CVC site | 1
  Grade 1-2 pain at right jugular Hohn catheter | 1
  Grade 1-2 injection site reaction (rash) | 1
  Grade 1-2 redness at Hohn catheter insertion site | 1
  Grade 1-2 right knee pain | 1
  Grade 1-2 diffuse pain | 1
  Grade 1-2 pain in leg | 1
  Grade 1-2 pain, skin nodule at biopsy site | 1
  Grade 1-2 transfusion reaction to packed red blood cells | 1
  Grade 1-2 chills | 1
  Grade 1-2 edema limbs | 1
  Grade 3-5 fatigue | 1
  Grade 1-2 fever | 3
  Grade 1-2 gait disturbance | 2
  Grade 1-2 injection site reaction | 8
  Grade 1-2 localized edema | 1
  Grade 1-2 malaise | 1
  Grade 1-2 non-cardiac chest pain | 2
  Grade 3-5 non-cardiac chest pain | 1
  Grade 1-2 allergic reaction | 3
  Grade 3-5 lung infection | 3
  Grade 3-5 sepsis | 2
  Grade 1-2 sinusitis | 1
  Grade 1-2 upper respiratory infection | 2
  Grade 1-2 urinary tract infection | 1
  Grade 3-5 urinary tract infection | 1
  Grade 1-2 bruising | 2
  Grade 1-2 fall | 3
  Grade 1-2 hip fracture | 1
  Grade 1-2 activated partial thromboplastin time prolonged | 2
  Grade 3-5 activated partial thromboplastin time prolonged | 1
  Grade 1-2 alanine aminotransferase increased | 3
  Grade 3-5 alanine aminotransferase increased | 1
  Grade 1-2 alkaline phosphatase | 5
  Grade 1-2 aspartate aminotransferase increased | 3
  Grade 3-5 aspartate aminotransferase increased | 2
  Grade 1-2 cardiac troponin T increased | 1
  Grade 1-2 creatinine increased | 4
  Grade 1-2 electrocardiogram QT corrected interval prolonged | 2
  Grade 3-5 electrocardiogram QT corrected interval prolonged | 1
  Grade 1-2 INR increased | 2
  Grade 1-2 serum amylase increased | 1
  Grade 1-2 weight gain | 1
  Grade 1-2 weight loss | 3
  Grade 1-2 anorexia | 6
  Grade 3-5 anorexia | 2
  Grade 1-2 dehydration | 1
  Grade 3-5 hyperglycemia | 1
  Grade 1-2 hyperuricemia | 2
  Grade 3-5 hyperuricemia | 1
  Grade 1-2 hypoalbuminemia | 5
  Grade 3-5 hypokalemia | 1
  Grades 3-5 hypomagmesemia | 1
  Grade 3-5 hypophosphatemia | 4
  Grade 3-5 tumor lysis syndrome | 1
  Grade 3-5 muscle weakness lower limb | 1
  Grade 1-2 neck pain | 1
  Grade 1-2 osteoporosis | 1
  Grade 1-2 pain in extremity | 1
  Grade 1-2 altered mental status | 1
  Grade 3-5 altered mental status | 1
  Grade 1-2 dizziness | 1
  Grade 1-2 headache | 3
  Grade 1-2 paresthesia | 2
  Grade 3-5 peripheral motor neuropathy | 1
  Grade 1-2 peripheral sensory neuropathy | 1
  Grade 1-2 somnolence | 1
  Grade 3-5 syncope | 1
  Grade 1-2 tremor | 2
  Grade 1-2 anxiety | 2
  Grade 1-2 confusion | 2
  Grade 1-2 depression | 2
  Grade 1-2 insomnia | 1
  Grade 1-2 hematuria | 3
  Grade 1-2 proteinuria | 1
  Grade 1-2 urinary incontinence | 1
  Grade 1-2 urinary retention | 2
  Grade 1-2 urinary tract pain | 1
  Grade 1-2 irregular menstruation | 1
  Grade 1-2 hemoptysis | 1
  Grade 1-2 atelectasis | 3
  Grade 1-2 dyspnea | 2
  Grade 3-5 dyspnea | 1
  Grade 1-2 hypoxia | 2
  Grade 3-5 hypoxia | 1
  Grade 1-2 nasal congestion | 1
  Grade 1-2 pleural effusion | 3
  Grade 1-2 productive cough | 1
  Grade 1-2 pulmonary edema | 2
  Grade 3-5 cellulitis | 1
  Grade 1-2 dry skin | 1
  Grade 1-2 erythema multiforme | 1
  Grade 1-2 pruritus | 2
  Grade 1-2 purpura | 3
  Grade 1-2 rash maculo-papular | 2
  Grade 1-2 scalp pain | 1
  Grade 1-2 hypertension | 4
  Grade 3-5 hypertension | 3
  Grade 1-2 hypotension | 2
  Grade 3-5 hypotension | 1

2. Secondary Outcome: Composite Complete Remission Rate (CRc=CR+CRi)
Description: Complete remission (CR) = an absolute neutrophil count (segs and bands) > 1,000/mcL, no circulating lymphoblasts, platelets ≥ 100,000/mcL; and < 5% marrow leukemia blast cells with complete disappearance of all measurable disease as confirmed by physical examination, CT scan and/or FDG-PET (Deauville criteria score of 1, 2, or 3)
  -Morphologic complete remission with incomplete blood count recovery (CRi)=Defined as CR with the exception of neutropenia < 1,000/mcL or thrombocytopenia <100,000/mcL
Time Frame: Completion of treatment (approximately 12 weeks)
Population: 2 participants were not evaluable for this outcome measure because they stopped treatment prior to disease response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: BL-8040 and Nelarabine
Number analyzed (Participants) | 10
Participants | 4

3. Secondary Outcome: Overall Response Rate (CR, CRi + PR)
Description: * Complete remission (CR) = an absolute neutrophil count (segs and bands) > 1,000/mcL, no circulating lymphoblasts, platelets ≥ 100,000/mcL; and < 5% marrow leukemia blast cells with complete disappearance of all measurable disease as confirmed by physical examination, CT scan and/or FDG-PET (Deauville criteria score of 1, 2, or 3)
  * Morphologic complete remission with incomplete blood count recovery (CRi)=Defined as CR with the exception of neutropenia < 1,000/mcL or thrombocytopenia <100,000/mcL
  * Partial remission (PR)=A PR requires all of the CR criteria except that marrow may still contain 5-25% leukemia blast cells. An absolute neutrophil count (segs and bands) ≥ 1000/mcL, no circulating blasts, and platelets > 100,000/mcL are requires as for a CR. For patients with measurable disease, a reduction of 50% or more in the sum of the products of the perpendicular diameters of all measurable lesions compared with pretreatment measurements and with no new or enlarging lesions
Time Frame: Through completion of treatment (median treatment length of 37.5 days, full range of 13-90 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: BL-8040 and Nelarabine
Number analyzed (Participants) | 10
Participants | 5

4. Secondary Outcome: Time to Response
Description: * Response is CR or CRi
  * Complete remission (CR) = an absolute neutrophil count (segs and bands) > 1,000/mcL, no circulating lymphoblasts, platelets ≥ 100,000/mcL; and < 5% marrow leukemia blast cells with complete disappearance of all measurable disease as confirmed by physical examination, CT scan and/or FDG-PET (Deauville criteria score of 1, 2, or 3)
  * Morphologic complete remission with incomplete blood count recovery (CRi)=Defined as CR with the exception of neutropenia < 1,000/mcL or thrombocytopenia <100,000/mcL
Time Frame: Through completion of treatment (median treatment length of 37.5 days, full range of 13-90 days)
Measure: Median (Full Range); unit: days
Arm/Group | Arm 1: BL-8040 and Nelarabine
Number analyzed (Participants) | 4
days | 20 [20 to 39]

5. Secondary Outcome: Duration of Response
Description: Defined as the interval from the date CR/CRi is documented to the date of recurrence or completion of follow-up if recurrence has not occurred.
Time Frame: Through date of recurrence or completion of follow-up (maximum of 2 years after completion of treatment)
Measure: Median (Full Range); unit: days
Arm/Group | Arm 1: BL-8040 and Nelarabine
Number analyzed (Participants) | 4
days | 280 [54 to 471]

6. Secondary Outcome: Event-free Survival (EFS)
Description: EFS is defined as the interval from the date of first dose of study drug to date of treatment failure, recurrence, of death due to any cause.
Time Frame: Through completion of follow-up (maximum of 2 years after completion of treatment)
Measure: Median (Full Range); unit: days
Arm/Group | Arm 1: BL-8040 and Nelarabine
Number analyzed (Participants) | 12
days | 23 [13 to 314]

7. Secondary Outcome: Overall Survival
Description: Defined as the date of first dose of study drug to the date of death from any cause.
Time Frame: Through completion of follow-up (maximum of 2 years after completion of treatment)
Measure: Median (Full Range); unit: days
Arm/Group | Arm 1: BL-8040 and Nelarabine
Number analyzed (Participants) | 12
days | 95 [24 to 440]

8. Secondary Outcome: Rate of Patients Who Proceed to alloHCT After Treatment
Description: Estimate rate of patients who proceed to alloHCT after treatment
Time Frame: Through completion of treatment (median treatment length of 37.5 days, full range of 13-90 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: BL-8040 and Nelarabine
Number analyzed (Participants) | 12
Participants | 3

9. Other Pre Specified Outcome: Interaction of Pretreatment Disease and White Blood Cell Count on Clinical Outcome
Description: Interaction of pretreatment disease and white blood cell count on clinical outcome
Time Frame: Up to 2 years after completion of treatment (approximately 116 weeks)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Interaction of Pretreatment Disease and Performance Status on Clinical Outcome
Description: Interaction of pretreatment disease and performance status on clinical outcome
Time Frame: Up to 2 years after completion of treatment (approximately 116 weeks)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Interaction of Pretreatment Disease and Immunophenotype on Clinical Outcome
Description: Interaction of pretreatment disease and immunophenotype on clinical outcome
Time Frame: Up to 2 years after completion of treatment (approximately 116 weeks)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Interaction of Pretreatment Disease and Cytogenetics on Clinical Outcome
Description: Interaction of pretreatment disease and cytogenetics on clinical outcome
Time Frame: Up to 2 years after completion of treatment (approximately 116 weeks)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Interaction of Pretreatment Disease and CXCR4 Expression on Lymphoblasts on Clinical Outcome
Description: Interaction of pretreatment disease and CXCR4 expression on lymphoblasts on clinical outcome
Time Frame: Up to 2 years after completion of treatment (approximately 116 weeks)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Interaction of Pretreatment Disease and Morphology on Clinical Outcome
Description: Interaction of pretreatment disease and morphology on clinical outcome
Time Frame: Up to 2 years after completion of treatment (approximately 116 weeks)
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Pharmacodynamic Effects of BL-8040 on T-lymphoblasts as Measured by Alterations in Lymphoblast Cell Cycle Status
Description: Pharmacodynamic effects of BL-8040 on T-lymphoblasts as measured by alterations in lymphoblast cell cycle status
Time Frame: Completion of treatment (approximately 12 weeks)
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Pharmacodynamic Effects of BL-8040 on T-lymphoblasts as Measured by Induction of Apoptosis in Lymphoblasts
Description: Pharmacodynamic effects of BL-8040 on T-lymphoblasts as measured by induction of apoptosis in lymphoblasts
Time Frame: Completion of treatment (approximately 12 weeks)
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Pharmacodynamic Effects of BL-8040 on T-lymphoblasts as Measured by Mobilization of Lymphoblasts Into the Peripheral Circulation
Description: Pharmacodynamic effects of BL-8040 on T-lymphoblasts as measured by mobilization of lymphoblasts into the peripheral circulation
Time Frame: Completion of treatment (approximately 12 weeks)
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Pharmacodynamic Effects of BL-8040 on T-lymphoblasts as Measured by Inhibition of CXCR4 Signaling on Lymphoblasts
Description: Pharmacodynamic effects of BL-8040 on T-lymphoblasts as measured by inhibition of CXCR4 signaling on lymphoblasts
Time Frame: Completion of treatment (approximately 12 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment through 30 days after the last study treatment (maximum of 4 cycles of treatment - each cycle is 21 days). All-cause mortality was collected from first dose of study treatment through completion of follow-up (maximum of 2 years following completion of treatment).
Arm/Group | Arm 1: BL-8040 and Nelarabine
All-Cause Mortality (participants affected / at risk) | 9/12
Serious Adverse Events (participants affected / at risk) | 8/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: BL-8040 and Nelarabine (N=12)
Leukocytosis (Blood and lymphatic system disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Fatigue (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Hip fracture (Injury, poisoning and procedural complications) | 1
Pain at BL-8040 injection site (Injury, poisoning and procedural complications) | 1
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered mental status (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: BL-8040 and Nelarabine (N=12)
Lymphadenopathy worsening (Blood and lymphatic system disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Infarct (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Chills (General disorders) | 1
Diffuse pain (General disorders) | 1
Edema limbs (General disorders) | 1
Fever (General disorders) | 3
Gait disturbance (General disorders) | 2
Injection site reaction (General disorders) | 8
Injection site reaction (rash) (General disorders) | 1
Localized edema (General disorders) | 1
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain at CVC site (General disorders) | 1
Pain in leg (General disorders) | 1
Transfusion reaction to pRBC (General disorders) | 1
"Feeling funny" post transfusion (General disorders) | 1
Allergic reaction (Immune system disorders) | 3
Lung infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Biopsy pain (Injury, poisoning and procedural complications) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Catheter pain, replacement (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Pain at right internal jugular Hohn catheter (Injury, poisoning and procedural complications) | 1
Pain, skin nodule at biopsy site (Injury, poisoning and procedural complications) | 1
Redness at Hohn catheter insertion site (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 5
Cardiac troponin T increased (Investigations) | 1
Creatinine increased (Investigations) | 4
Electrocardiogram QT corrected interval prolonged (Investigations) | 3
INR increased (Investigations) | 2
Serum amylase increased (Investigations) | 1
Weight gain (Investigations) | 1
Weight loss (Investigations) | 3
White blood cell count increased post BL-8040 injection (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Right knee pain (Musculoskeletal and connective tissue disorders) | 1
Altered mental status (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Paresthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Urinary tract pain (Renal and urinary disorders) | 1
Irregular menstruation (Renal and urinary disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2
Cellulitis on hand (Infections and infestations) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Purpura (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT02763384/Prot_SAP_000.pdf